CLINICAL TRIAL: NCT03690661
Title: Using Serious Games to Improve Social Skills in Autism
Acronym: SAGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, K. Suzanne Scherf, Associate Professor of Psychology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R33MH110624 (NIH); R33MH110624 (NIH)
Record Dates: First submitted 2018-09-20; First posted 2018-10-01 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: adolescent; face; social skills; video game
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Facies; Social Skills

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Video Game (Experimental): Participants will play the Intervention Video Game for 3 months, 3 times a week for a minimum of 30 minutes each session
  Interventions: Behavioral: Intervention Video Game
- Control Video Game (Placebo Comparator): Participants will play the Control Video Game for 3 months, 3 times a week for a minimum of 30 minutes each session
  Interventions: Behavioral: Placebo Control Game

INTERVENTIONS:
Behavioral: Intervention Video Game — The intervention game employs evidence-based "serious game" mechanics (e.g., storylines, long-term goals, scaling difficulty) to design a learning environment that maximizes opportunities for adolescents with ASD to discover the functional utility of eye gaze cues.
  Arms: Intervention Video Game
Behavioral: Placebo Control Game — The placebo game will have all the elements of the serious game mechanics of the intervention game (narrative storylines, long-term goals, scaling difficulty), but will not provide the learning opportunities regarding eye gaze cues.
  Arms: Control Video Game

SUMMARY:
The investigators will conduct a small-scale randomized control trial comparing the intervention game to an active control game, and will assess outcomes at multiple time points (pre-, post-, 6-month follow-up). These outcomes will include a wide range of behaviors that are measured along a continuum from controlled lab-based tasks to uncontrolled, real-world social interactions between dyads.

DETAILED DESCRIPTION:
The investigators will conduct a small-scale randomized control trial comparing the intervention game to an placebo control game, and will assess outcomes at multiple time points (pre-, post-, 6-month follow-up). These outcomes will include a wide range of behaviors that are measured along a continuum from controlled lab-based tasks to real-world social interactions between dyads. The aims are evaluating 1) changes in the target mechanisms (social attention to faces, sensitivity to eye gaze cues) for the intervention relative to active control group, 2) engagement of intermediate mechanisms, including face-processing behaviors and real-world social communication behaviors, and 3) the relation between engagement of the target and intermediate mechanisms and symptom outcomes. Evidence of changes in autism social symptoms resulting from changing visual attention to faces and/or improved ability to understand eye gaze cues will provide clear evidence to inform a "go" decision about the therapeutic target for further clinical development.

ELIGIBILITY:
Inclusion Criteria:

1. parent/caregiver of an adolescent with a diagnosis of autism spectrum disorder (ASD),
2. parent/caregiver and adolescent with ASD both native English speakers,
3. adolescent with ASD aged between 10-18 years at pre-test,
4. adolescent has normal vision and hearing with correction as reported by caregiver,
5. adolescent is able to use a computer for the purposes of game play,
6. adolescent scores < 80% correct (i.e., 0.5 SD less than Mean of typically developing adolescents) on online eye gaze screening task,
7. ASD diagnosis of adolescent confirmed via Parent-report SCQ and clinical interview with adolescent to assess DSM-V criteria (borderline cases also undergo ADI interview);
8. Full Scale IQ of adolescent determined to be between 70-130;
9. reading ability of adolescent determined to be at least a 2nd grade level;
10. adolescent is capable of cooperating with testing;
11. parent/caregiver and adolescent both consent/assent to participate in the research.

Exclusion Criteria:

1. having seizures within the previous two years
2. no stable internet connection in the home
3. refusing to consent/assent to take part in the research
4. 18 and have a legal guardian, which prohibits them from legally consenting for themselves
5. 18 and cannot understand the consent as indicated by failing a quiz prior to signing the consent.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Primary Target Eye Gaze Mechanisms - Performance Accuracy | 6 months
  Performance accuracy will be acquired from both a static and a dynamic task of eye gaze cue following, which will be analyzed separately (ie 6 months from pre-intervention).
Primary Target Eye Gaze Mechanisms - Visual Fixation | 6 months
  Eye tracking measures of visual fixation will be acquired in both a static and a dynamic task of eye gaze cue following, which will be analyzed separately (ie 6 months from pre-intervention).
Social Symptoms - Social Skills Inventory System (SSIS) | 6 months
  Social skills and problematic behaviors will be assessed via parent- and self-reported responses on the SSIS. These measures will be administered at multiple time points including pre-intervention, post-intervention, and 3 months after the intervention (ie 6 months from pre-intervention).
Autism Behaviors - Social Responsiveness Scale 2nd Edition (SRS-2) | 6 months
  To assess potential changes in autism-like behaviors and symptoms, parents will complete the SRS-2 at each of 3 time points (pre-intervention, post-intervention, 3-month follow-up after intervention completion).

SECONDARY OUTCOMES:
Intermediate Face Processing Mechanisms - Face Identity (CFMT) | 6 months
  Accuracy in face recognition will be assessed via standardized measures including Cambridge face memory task (CFMT) at each time point including pre-intervention, post-intervention, and 3 months after the intervention (ie 6 months from pre-intervention).
Intermediate Face Processing Mechanisms - Object Identity (CBMT) | 6 months
  Accuracy in object recognition will be assessed via standardized measures including Cambridge bike memory task (CBMT) at each time point including pre-intervention, post-intervention, and 3 months after the intervention (ie 6 months from pre-intervention).
Intermediate Face Processing Mechanisms - Face Expression Identification - (CAM) | 6 months
  Accuracy in face expression identification will be assessed via standardized measures including the face portion of the Cambridge Affective Memory task (CAM) at each time point including pre-intervention, post-intervention, and 3 months after the intervention (ie 6 months from pre-intervention).
Intermediate Face Processing Mechanisms - Face Expression Identification - (RMET) | 6 months
  Accuracy in face expression identification will be assessed via standardized measures including the face portion of the Reading the Mind in the Eyes Test (RMET) at each time point including pre-intervention, post-intervention, and 3 months after the intervention (ie 6 months from pre-intervention).
Face-to-Face Social Interactions - Visual Fixations | 6 months
  Eye tracking measures (ie visual fixations) will be collected during a naturalistic social conversation. Additionally, eye tracking measures will be collected during an interactive cued eye gaze task, which requires participants to select the object that a real person is looking at. These measures will be assessed at multiple time points including pre-intervention, post-intervention, and 3 months after the intervention (ie 6 months from pre-intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Suzy Scherf, Principal Investigator — Penn State University
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants will be invited to share de-identified data acquired from this study with the National Institutes of Health Data Archive
Supporting Information: Study Protocol, ICF